CLINICAL TRIAL: NCT04858503
Title: An Internet-based Cardiac Rehabilitation Enhancement (i-CARE) Intervention to Support Self-care of Patients With Coronary Artery Disease: A Mixed-method Study
Brief Title: An Internet-based Cardiac Rehabilitation Enhancement (i-CARE) Intervention to Support Self-care of Patients With Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Polly Wai-Chi Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NTWC/REC/20139
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: Self-care; Model of care; Mobile app; Empowerment; Nurse-led; Disease Management; Risk factor control
MeSH Terms: conditions — Coronary Artery Disease; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internet-based cardiac rehabilitation enhancement intervention (Experimental): internet-based cardiac rehabilitation enhancement intervention
  Interventions: Other: internet-based cardiac rehabilitation enhancement intervention
- conventional cares as arranged by hospital or community centers (No Intervention): Participants will receive conventional cares as arranged by hospital or community centers

INTERVENTIONS:
Other: internet-based cardiac rehabilitation enhancement intervention — Participants in the intervention group will receive a 12-week i-CARE intervention, which will be designed to cover the core elements of CAD self-care: self-care maintenance, self-care monitoring and self-care management. The intervention will comprise: 1) a single individualized face-to-face session and 2) an internet-based intervention through a mobile application. Various behaviour change techniques will be used to increase the self-efficacy of CAD patients in enacting self-care behaviours.
  Arms: internet-based cardiac rehabilitation enhancement intervention

SUMMARY:
This study aims to examine the effects of an internet-based cardica rehabilitation enhancement (i-CARE) programme for coronary artery disease (CAD) patients on self-care behaviour, biomarkers, physiological, anthropometric parameters, clinical outcomes and self-reported health outcomes and to understand why and how i-CARE influences patients' health behaviours.

DETAILED DESCRIPTION:
This study aims to examine the effects of an internet-based cardica rehabilitation enhancement (i-CARE) programme for coronary artery disease (CAD) patients on self-care behaviour, biomarkers, physiological, anthropometric parameters, clinical outcomes and self-reported health outcomes and to understand why and how i-CARE influences patients' health behaviours.

Cardiovascular disease, a highly prevalent morbidity, is the number one cause of death worldwide and has become a significant public health concern. The majority of these deaths are attributed to an acute manifestation of coronary artery disease (CAD), defined as a narrowing of the coronary arteries that causes insufficient myocardial blood flow. CAD has reached an unequivocal pandemic status globally and locally. CAD imposes not only significant physical and psychosocial burdens on patients, but also enormous service demands on healthcare systems.As a chronic condition, CAD requires patients to practice persistent self-care in a long-term manner for successful disease management. Self-care is considered fundamental to the prevention and management of chronic diseases. Yet, a significant proportion of the CAD population is still engaging in full-time employment, their time availability restricts them to participate in traditional health promotional activities. According to recent systematic reviews, substantial evidence has accumulated to support the positive effects of internet-delivered interventions. Therefore, an internet-based approach with self-care cardiac rehabilitation enhancement may be ab better method of engaging patients in the learning process and arousing their inherent capacities to maintain behavioral modifications. This mixed-method study consists of a two-arm randomized controlled trial and an exploratory qualitative study. For the randomized controlled trial plans to recruit 268 adults from Queen Mary Hospital and Care for Your Heart. Eligible participants will be CAD patients who aged 18 above, living in the community, owning a smartphone with internet access, communicable in Cantonese and able to type in Chinese or English. The participants will be randomly allocated to the intervention or control group to receive i-CARE or usual care, respectively. The study hypotheizes that the CAD patients who receive the i-CARE intervention will report better changes in self-care behaviours, blood pressure, cholesterols, waist-to-height ratio, functional status and HRQoL at 3 and 6 months after the intervention, than those who receive usual care and that the CAD patients who receive the i-CARE intervention will report fewer cardiovascular event rates and mortality at 6 months after the intervention, than those who receive usual care. The findings will advance our knowledge of the empirical effects of internet-based cardiac rehabilitation programme on CAD patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* living in the community,
* own a smartphone with internet access,
* communicable in Cantonese,
* type in Chinese or English,
* with a confirmed diagnosis of CAD.

Exclusion Criteria:

* enrolled to a structured centre-based or home-based cardiac rehabilitation program, (2) psychiatric problems,
* impaired cognitive functioning (i.e. Abbreviated Mental Test ≤6), and
* terminal disease with life expectancy < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-care behaviour | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  the Chinese version of Self-Care of Coronary Heart Disease Inventory (SC-CHDI). This self-reported SC-CHDI (22 items) measures self-care maintenance, self-care management and self-care confidence on a four-point response scale. Each subscale score is transformed to 100 points, with higher scores indicate better self-care for that attribute.

SECONDARY OUTCOMES:
Biomarkers: lipid profile | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  POCT
Physiological: blood pressure | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  Measure both systolic and diastolic blood pressure
Anthropometric: waist-to-height ratio | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  Measure waist-to-height ratio
Clinical: Cardiovascular event rates and mortality | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  the admissions, cardiovascular event rates and mortality data will be retrieved
Self-reported health outcomes: functional status | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  The functional status will be measured with the Chinese version of Seattle Angina Questionnaire. This 19-item questionnaire consists of five subscales, including physical limitation, angina stability, angina frequency, treatment satisfaction and the disease perception. The respondents have to rate on a 1 to 5 or 6 sequentially coded status. The subscale scores are transformed to a scale of 0 to 100, with higher scores indicate higher level of functioning/ satisfaction and fewer limitations.
Health-related Quality of life (HRQoL) | Change from Baseline at the 3 months (after the intervention) and 6 months (follow up)
  The Chinese version of MacNew will be used to measure disease-specific HRQoL.22 It consists of 27 items measuring HRQoL in three domains (physical, emotional and social). Each item is rated on a 1-7 scale, and a global score is calculated by summing the item scores, a higher score represents better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Li, Dr, Principal Investigator — The University of Hong Kong, School of Nursing
Locations (1):
- The School of Nursing, Hong Kong, Hong Kong

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04858503/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT04858503/ICF_002.pdf